CLINICAL TRIAL: NCT06183619
Title: Superior Vena Cava Isolation Plus Pulmonary Vein Isolation for Paroxysmal Atrial: a Multi-center Retrospective Study
Brief Title: Superior Vena Cava Isolation Plus Pulmonary Vein Isolation for Paroxysmal Atrial Fibrillation
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jun Liu,MD, Attending doctor, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: T2020-ZX019
Record Dates: First submitted 2023-12-14; First posted 2023-12-27 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary vein isolation plus superior vena cava isolation
  Interventions: Procedure: Pulmonary vein isolation plus superior vena cava isolation
- Pulmonary vein isolation
  Interventions: Procedure: Pulmonary vein isolation

INTERVENTIONS:
Procedure: Pulmonary vein isolation plus superior vena cava isolation — Pulmonary vein isolation plus superior vena cava isolation
  Groups: Pulmonary vein isolation plus superior vena cava isolation
Procedure: Pulmonary vein isolation — Pulmonary vein isolation only
  Groups: Pulmonary vein isolation

SUMMARY:
Pulmonary vein isolation (PVI) for paroxysmal atrial fibrillation (PAF) has limited success. The superior vena cava (SVC) has been identified as one of the most common non-pulmonary vein triggers for PAF. It is estimated that SVC isolation (SVCI) could improve the clinical results of patients with PAF. However, results from previous studies about SVCI remain controversial. Safety concerns for SVCI may outweigh its benefits and lead to inadequate ablation. To address this issue, the introduction of a quantitative ablation index (AI) for SVCI may provide a solution. Therefore, the investigators sought to initiate a retrospective, multi-center study, to explore the efficacy and safety of quantitative SVCI in addition to PVI in PAF.

DETAILED DESCRIPTION:
Catheter ablation has emerged as an effective treatment for drug-refractory PAF and is recommended as first-line therapy by current guidelines. PVI is considered the cornerstone of catheter ablation for atrial fibrillation (AF). However, despite persistent PVI, a subgroup of patients may experience recurrent AF due to focal ectopic discharges originating outside the pulmonary veins. Among the non-pulmonary vein triggers, the SVC stands out as a common culprit, making it a promising ablation target for maintaining sinus rhythm. Nevertheless, results from previous studies that evaluated the efficacy of SVCI showed conflicting results. One possible explanation is that SVC is adjacent to critical anatomical structures (such as the sinus node and the phrenic nerve), which raises safety concerns and often leads to inadequate ablation.

Therefore, it is necessary to establish a standardized ablation procedure for SVCI, ensuring both safety and efficacy. To address this issue, the investigators proposed the concept of "quantitative ablation for SVCI." By introducing AI as a quantitative measure, it is possible to achieve precise catheter ablation while minimizing the risk of procedure-related complications.

This study aimed to investigate the safety and feasibility of quantitative AI-guided SVCI in addition to PVI. Participants with PAF who required catheter ablation will be consecutively enrolled in three hospitals in China.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic paroxysmal AF that are unresponsive to antiarrhythmic drugs (one or more than one).
* Willing to undergo catheter ablation for AF.

Exclusion Criteria:

* History of any type of catheter ablation for cardiac arrhythmias.
* Sinus node dysfunction that requires permanent pacemaker implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic paroxysmal AF that are unresponsive to antiarrhythmic drugs (one or more than one).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
AT/AF recurrence | 12 months
  atrial fibrillation, atrial flutter, atrial tachycardia over 30s

CONTACTS AND LOCATIONS:
Overall Officials: Jun Liu, MD, PhD, Principal Investigator — Fuwai hospital, Chinese Academy of Medical Science
Locations (1):
- Chinese Academy of Medical Science, Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No